CLINICAL TRIAL: NCT00907504
Title: Randomized, Open Label, Phase 3 Clinical Study To Evaluate The Effect Of The Addition Of CP-751,871 To Gemcitabine And Cisplatin In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Study Of The Effect Of CP-751,871 In Combination With Gemcitabine And Cisplatin In Patients With Advanced Non-Small Cell Lung Cancer
Acronym: ADVIGO1017
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4021017
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — figitumumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CP-751,871 + Gemcitabine + Cisplatin (Experimental): investigational arm
  Interventions: Drug: CP-751,871; Drug: Cisplatin; Drug: Gemcitabine
- Gemcitabine + Cisplatin (Active Comparator): standard of care
  Interventions: Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 20mg/kg every 3 weeks
  Arms: CP-751,871 + Gemcitabine + Cisplatin
Drug: Cisplatin — Cisplatin 80 mg/m2 every 3 weeks
  Arms: CP-751,871 + Gemcitabine + Cisplatin
Drug: Gemcitabine — Gemcitabine 1,250 mg/m2 Day1+8 of evey 3 week-cycle
  Arms: CP-751,871 + Gemcitabine + Cisplatin
Drug: Cisplatin — Cisplatin 80 mg/m2 every 3 weeks
  Arms: Gemcitabine + Cisplatin
Drug: Gemcitabine — Gemcitabine 1,250 mg/m2 Day1+8 of evey 3 week-cycle
  Arms: Gemcitabine + Cisplatin

SUMMARY:
Gemcitabine and cisplatin given together is a standard treatment option for advanced lung cancer patients. The purpose of this study is to assess if the life span is longer in patients taking the investigational drug CP-751,871 in combination with gemcitabine and cisplatin compared to gemcitabine and cisplatin alone. Considering a 10% rate of drop-outs, 1,210 participants will be required in order to have an adequate sample size (1,100 evaluable patients) and power to detect a 30% prolongation of survival on the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Non-Small Cell Lung Cancer (NSCLC), advanced, chemotherapy-naive
* Male or female > 18 years
* Eastern Oncology Cooperative Group (ECOG) Performance Status (PS) 0 or 1
* Adequate organ function

Exclusion Criteria:

* Uncontrolled hypertension or diabetes;
* Pregnant female;
* Symptomatic Central Nervous System (CNS) metastasis, requirement for chronic corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Dec 2012

SECONDARY OUTCOMES:
Progression Free survival | Dec 2011
Objective Response | Dec 2011
Overall Safety Profile | Dec 2012
Patient Reported Outcome | Dec 2012
Pharmacokinetics | Dec 2012
Anti-drug Antibody | Dec 2012
Biomarker Analysis | Dec 2012

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4021017&StudyName=Study%20Of%20The%20Effect%20Of%20CP-751%2C871%20In%20Combination%20With%20Gemcitabine%20And%20Cisplatin%20In%20Patients%20With%20Advanced%20Non-Small%20Cell%20Lung%20Cancer